CLINICAL TRIAL: NCT06829485
Title: Florida Community-Engaged Research Alliance (FL-CEAL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Westat (Other)
Responsible Party: Principal Investigator, Olveen Carrasquillo, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20240463; OT2HL158287 (NIH); 6922-03-COVID-S005 (Other Grant/Funding Number: Westat)
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Health, Subjective
Keywords: Health Determinants
MeSH Terms: interventions — Community Health Workers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health worker Group (Experimental): Participants in this group will be linked to a community health worker for up to 6 months and also be offered the opportunity to participate in group level activities
  Interventions: Behavioral: Community health workers (CHW)
- Educational material group (Active Comparator): Participants in this group will be provided with educational material on health resources for up to 6 months
  Interventions: Behavioral: Educational Materials

INTERVENTIONS:
Behavioral: Community health workers (CHW) — Participants will meet with a Community Health Worker (CHW) who will help facilitate and provide personalized navigation to existing resources for addressing health challenges such as food insecurity and access to care. CHW will meet with participants in person or virtually at least three times for approximately 15-60 minutes for over the six month period
  Arms: Community Health worker Group
Behavioral: Educational Materials — Participants will receive one time educational materials including information of existing health resources. Participants will be able to review materials at participant discretion.
  Arms: Educational material group

SUMMARY:
The purpose of the study is learn more about ways to help people with non-medical issues that can affect participant health. The study team will examine if Community Health Workers, members of a community who provide basic health and medical care within communities, are more helpful to people with non-medical issues than simple reading materials on how participants can do it themselves.

ELIGIBILITY:
Inclusion Criteria:

* Individuals living within the target community who do not plan to move out of the community within the next six months
* Having two un-met SDOH needs

Site Specific Inclusion Criteria:

University of Miami/ Healthy Little Havana Inclusion Criteria

* Age 18 and over

Health Choice Network/ Broward Community Health Center/ Genesis Community Health Center Inclusion Criteria

* Age 18 and over

Florida International University Inclusion Criteria -Latina Women Age 18 and over

Mayo Clinic Florida Inclusion Criteria

-Age 21 and over

Florida A&M University/ Mother Care Network Inclusion Criteria

* Female minors between the ages 11-14 years
* Black/African American; Hispanic or Non-Hispanic ethnicity

University of Florida Inclusion Criteria

* Women aged 18 and over
* Pregnant and recently post-partum minority women

Exclusion Criteria:

* Are unable or unwilling to consent
* Plans to move out of the community during the next six months
* Enrollment in a research study addressing Social Determinants Determinants Of Health (SDOH) in the last three years.
* Prisoners

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in General well-being (GWB), measured by the Personal Wellbeing Index (PWI) | Baseline, 6 months
  In the PWI, each item is rated on a 0-to-10 scale (0 = No satisfaction at all; 10 = Very satisfied).

SECONDARY OUTCOMES:
Change in number of participants health insurance status as measured by CEAL Common Survey 4 (CS4) | Baseline, 6 months
  Health insurance status will measured by the number of participants who answered yes to the health insurance status
Change in number of participants having a usual source of care as measured by CEAL Common Survey 4 (CS4) | Baseline, 6 months
  Having a usual source of care will measured by the number of participants who answered yes to having usual source of care
Change in number of participants delayed medical care as measured by CEAL Common Survey 4 (CS4) | Baseline, 6 months
  Delayed medical care will measured by the number of participants who answered yes to having delayed medical care due the cost.
Food Insecurity as measured by U.S. Department of Agriculture Economic Research Service Questionnaire | Baseline, 6 months
  Food security status is assigned as follows:
  Raw score 0-1-High or marginal food security (raw score 1 may be considered marginal food security, but a large proportion of households that would be measured as having marginal food security using the household or adult scale will have raw score zero on the six-item scale) Raw score 2-4-Low food security Raw score 5-6-Very low food security

CONTACTS AND LOCATIONS:
Overall Officials: Olveen Carrasquillo, MD, Principal Investigator — University of Miami
Locations (7):
- United States (7):
  - University of Florida, Gainesville, Florida
  - Mayo Clinic Florida Comprehensive Cancer Center, Jacksonville, Florida
  - Healthy Little Havana, Miami, Florida
  - Florida International University, Miami, Florida
  - University of Miami, Miami, Florida
  - Health Choice Network, Miami, Florida
  - Florida A&M University, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: No